CLINICAL TRIAL: NCT00452530
Title: A Phase 3, Randomized, Double-blind, Active-controlled (Enoxaparin 40 mg QD), Parallel-group, Multi-center Study to Evaluate the Safety and Efficacy of Apixaban in Subjects Undergoing Elective Total Knee Replacement Surgery (The ADVANCE - 2 Study)
Brief Title: Study of an Investigational Drug for the Prevention of Thrombosis-related Events Following Knee Replacement Surgery
Acronym: ADVANCE-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV185-047; EUdraCT: 2006-006896-19
Record Dates: First submitted 2007-03-23; First posted 2007-03-27 (Estimated); Results first posted 2014-05-13 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism
Keywords: Prevention of deep vein thrombosis and pulmonary embolism after total knee replacement surgery
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — Enoxaparin; apixaban

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apixaban, 2.5 mg BID + Placebo (Experimental): Participants received apixaban, 2.5-mg tablets twice daily (BID), plus a matching enoxaparin-placebo injection 12 (±3) hours prior to hip-replacement surgery through 11 (±2) days after the day of surgery.
  Interventions: Drug: Apixaban; Drug: Enoxaparin-matching placebo
- Enoxaparin, 40 mg QD + Placebo (Active Comparator): Participants received enoxaparin, 40-mg subcutaneous injection once daily (QD), plus a matching apixaban-placebo tablet 12 (±3) hours prior to hip-replacement surgery through 11 (±2) days after the day of surgery.
  Interventions: Drug: Enoxaparin; Drug: Apixaban-matching placebo

INTERVENTIONS:
Drug: Enoxaparin — 40 mg, administered once daily by subcutaneous injection, for 12 days
  Other Names: Lovenox®
  Arms: Enoxaparin, 40 mg QD + Placebo
Drug: Apixaban — 2.5 mg, administered twice daily as tablets, for 12 days
  Other Names: BMS-562247
  Arms: Apixaban, 2.5 mg BID + Placebo
Drug: Enoxaparin-matching placebo — Administered once daily by subcutaneous injection
  Arms: Apixaban, 2.5 mg BID + Placebo
Drug: Apixaban-matching placebo — Oral tablet administered twice daily
  Arms: Enoxaparin, 40 mg QD + Placebo

SUMMARY:
The purpose of this study is to learn whether apixaban prevents the development of blood clots in the leg (deep vein thrombosis) and lung (pulmonary embolism), which sometimes occur after knee replacement surgery, and to compare the efficacy of apixaban with that of enoxaparin (Lovenox®) in the prevention of these clots. The safety of apixaban will also be studied.

ELIGIBILITY:
Key Inclusion Criteria

* Patients scheduled for either elective unilateral or same-day bilateral total knee replacement surgery (TKR) or a revision of at least 1 component of a TKR
* Patients willing and able to undergo bilateral ascending contrast venography

Key Exclusion Criteria

* Known or suspected hereditary or acquired bleeding or coagulation disorders in the participant or his or her first-degree relative
* Known or suspected history of heparin-induced thrombocytopenia
* Known coagulopathy
* Active bleeding or at high risk for bleeding
* Brain, spinal, ophthalmologic, or major surgery or trauma within the past 90 days
* Active hepatobiliary disease
* Alcohol and/or substance abuse within the past year
* Any condition for which, in the opinion of the investigator, surgery or administration of an anticoagulant was contraindicated
* Two consecutive blood pressure readings within 15 to 30 minutes with supine systolic blood pressure >180 mm Hg or supine diastolic blood pressure >105 mm Hg
* Clinically significant laboratory abnormalities at the enrollment visit:

  * Hemoglobin <10 g/dL
  * Platelet count <100,000/mm^3
  * Creatinine clearance <30 mL/min, as estimated by the method of Cockcroft and Gault
  * Alanine aminotransferase or aspartate aminotransferase level >2*upper limit of normal (ULN) or a total bilirubin ≥1.5*ULN (unless an alternative causative factor such as Gilbert's syndrome was identified)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3221 (Actual)
Dates: Start 2007-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (102):
- Austria (6):
  - Local Institution, Graz
  - Local Institution, Innsbruck
  - Local Institution, Linz
  - Local Institution, Vienna
  - Local Institution, Wels
  - Local Institution, Wiener Neustadt
- Belgium (2):
  - Local Institution, Antwerp
  - Local Institution, Hasselt
- Brazil (2):
  - Local Institution, Belo Horizonte - Mg, Minas Gerais
  - Local Institution, São Paulo, São Paulo
- Local Institution, Santiago, Santiago Metropolitan, Chile
- China (3):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Qingdao, Shandong
  - Local Institution, Shanghai, Shanghai Municipality
- Colombia (3):
  - Local Institution, Bogotá
  - Local Institution, Cali
  - Local Institution, Medellín
- Czechia (5):
  - Local Institution, Brno
  - Local Institution, Chomutov
  - Local Institution, Pardubice
  - Local Institution, Prague
  - Local Institution, Uherské Hradiště
- Denmark (4):
  - Local Institution, Hellerup
  - Local Institution, Hvidovre
  - Local Institution, Kolding
  - Local Institution, Viborg
- France (4):
  - Local Institution, Monaco
  - Local Institution, Nice
  - Local Institution, Paris
  - Local Institution, Saint-Saulve
- Germany (10):
  - Local Institution, Bad Mergentheim
  - Local Institution, Bochum
  - Local Institution, Brandenburg
  - Local Institution, Dresden
  - Local Institution, Frankfurt
  - Local Institution, Frankfurt am Main
  - Local Institution, Halle/S
  - Local Institution, Kremmen Ot Sommerfeld
  - Local Institution, Rheinfelden
  - Local Institution, Witten
- Hungary (2):
  - Local Institution, Szeged
  - Local Institution, Szekszárd
- India (5):
  - Local Institution, Ahmedabad, Gujarat
  - Local Institution, Ludhiana, Punjab
  - Local Institution, Bangalore
  - Local Institution, Baroda
  - Local Institution, Mangalore
- Israel (5):
  - Local Institution, Jeruselem
  - Local Institution, Petah Tikva
  - Local Institution, Safed
  - Local Institution, Tel Aviv
  - Local Institution, Tel Litwinsky
- Italy (5):
  - Local Institution, Abano Terme (Pd)
  - Local Institution, Bologna
  - Local Institution, Pordenone
  - Local Institution, Roma
  - Local Institution, San Donato Milanese (Mi)
- Local Institution, Kuala Lumpur, Kuala Lumpur, Malaysia
- Mexico (5):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Zapopan, Jalisco
  - Local Institution, San Luis Potosí City, San Luis Potosí
  - Local Institution, Hermosillo, Sonora
  - Local Institution, Veracruz, Veracruz
- Norway (3):
  - Local Institution, Ålesund
  - Local Institution, Gjettum
  - Local Institution, Kongsvinger
- Philippines (2):
  - Local Institution, Manila
  - Local Institution, Quezon City
- Poland (4):
  - Local Institution, Bytom
  - Local Institution, Gdansk
  - Local Institution, Warsaw
  - Local Institution, Wroclaw
- Russia (7):
  - Local Institution, Chelyabinsk
  - Local Institution, Kazan'
  - Local Institution, Lipetsk
  - Local Institution, Moscow
  - Local Institution, Rostov-on-Don
  - Local Institution, Saint Petersburg
  - Local Institution, Samara
- Local Institution, Singapore, Singapore
- South Africa (6):
  - Local Institution, Randburg, Free State
  - Local Institution, Johannesburg, Gauteng
  - Local Institution, Pretoria, Gauteng
  - Local Institution, Somerset West, Western Cape
  - Local Institution, Tygerberg, Western Cape
  - Local Institution, Worcester, Western Cape
- South Korea (2):
  - Local Institution, Jeonnam
  - Local Institution, Seoul
- Spain (5):
  - Local Institution, Badalona-Barcelona
  - Local Institution, Barcelona
  - Local Institution, Madrid
  - Local Institution, Santiago de Compostela
  - Local Institution, Valencia
- Local Institution, Borås, Sweden
- Ukraine (6):
  - Local Institution, Cherkassy
  - Local Institution, Chernivtsy
  - Local Institution, Dnipropetrovsk
  - Local Institution, Ivano-Frankivsk
  - Local Institution, Kyiv
  - Local Institution, Sevastopol
- United Kingdom (2):
  - Local Institution, London, Greater London
  - Local Institution, Epsom, Surrey

REFERENCES:
- [Derived] Jamieson MJ, Byon W, Dettloff RW, Crawford M, Gargalovic PS, Merali SJ, Onorato J, Quintero AJ, Russ C. Apixaban Use in Obese Patients: A Review of the Pharmacokinetic, Interventional, and Observational Study Data. Am J Cardiovasc Drugs. 2022 Nov;22(6):615-631. doi: 10.1007/s40256-022-00524-x. Epub 2022 May 16. PMID 35570249
- [Derived] Pineo GF, Gallus AS, Raskob GE, Chen D, Ramirez LM, Ramacciotti E, Lassen MR, Wang L. Apixaban after hip or knee arthroplasty versus enoxaparin: efficacy and safety in key clinical subgroups. J Thromb Haemost. 2013 Mar;11(3):444-51. doi: 10.1111/jth.12109. PMID 23279103
- [Derived] Lassen MR, Raskob GE, Gallus A, Pineo G, Chen D, Hornick P; ADVANCE-2 investigators. Apixaban versus enoxaparin for thromboprophylaxis after knee replacement (ADVANCE-2): a randomised double-blind trial. Lancet. 2010 Mar 6;375(9717):807-15. doi: 10.1016/S0140-6736(09)62125-5. PMID 20206776
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 3221 patients enrolled, 3057 were randomized. Primary participants=those who were randomized and had an adjudicated evaluable bilateral venogram or an adjudicated venous thromboembolic event or died. Evaluable participants=those with significant protocol deviations expected to affect the primary endpoint.
Groups:
- Apixaban, 2.5 mg BID + Placebo: Participants received apixaban, 2.5 mg twice daily (BID), as oral tablets, and matching enoxaparin-placebo injection once daily (QD)
- Enoxaparin, 40 mg QD + Placebo: Participants received enoxaparin, 40 mg QD subcutaneously, and matching apixaban-placebo tablets BID
Period: Overall Study
Arm/Group | Apixaban, 2.5 mg BID + Placebo | Enoxaparin, 40 mg QD + Placebo
Started | 1528 (Randomized) | 1529 (Randomized)
Received Treatment | 1501 | 1508
Evaluable Participants | 907 | 921
Primary Participants | 976 | 997
Completed | 1392 | 1393
Not Completed | 136 | 136
Not completed — Death | 1 | 0
Not completed — Adverse Event | 40 | 44
Not completed — Withdrawal by Subject | 68 | 57
Not completed — Lost to Follow-up | 1 | 0
Not completed — Poor compliance/noncompliance | 1 | 2
Not completed — No longer met study criteria | 18 | 22
Not completed — Other | 7 | 11

BASELINE CHARACTERISTICS:
Population: All participants randomized to treatment
Groups:
- Total: Total of all reporting groups
Arm/Group | Apixaban, 2.5 mg BID + Placebo | Enoxaparin, 40 mg QD + Placebo | Total
Number analyzed (Participants) | 1528 | 1529 | 3057
Age, Continuous [Median (Standard Deviation); unit: Years] | 67 (9.85) | 67 (9.82) | 67 (9.84)
Age, Customized [Number; unit: Participants]
  Younger than 65 years | 632 | 636 | 1268
  65 years to younger than 75 years | 608 | 576 | 1184
  75 years and older | 288 | 317 | 605
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1089 | 1127 | 2216
  Male | 439 | 402 | 841
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 1216 | 1211 | 2427
  Black/African American | 14 | 17 | 31
  Asian | 252 | 254 | 506
  Native Hawaiian/Other Pacific Islander | 1 | 1 | 2
  Other [Not specified] | 45 | 46 | 91
  Hispanic/Latino | 0 | 1 | 1
  Not Hispanic/Latino | 53 | 57 | 110
  Ethnicity not reported | 1475 | 1471 | 2946
Region of Enrollment [Number; unit: Participants]
  Philippines | 12 | 14 | 26
  Spain | 61 | 60 | 121
  Ukraine | 181 | 182 | 363
  Russian Federation | 150 | 156 | 306
  Israel | 43 | 43 | 86
  Chile | 1 | 5 | 6
  Colombia | 36 | 35 | 71
  Italy | 69 | 69 | 138
  India | 92 | 92 | 184
  France | 72 | 68 | 140
  Malaysia | 4 | 4 | 8
  Denmark | 26 | 23 | 49
  South Africa | 56 | 56 | 112
  China | 90 | 90 | 180
  Korea, Republic of | 40 | 38 | 78
  Austria | 156 | 151 | 307
  United Kingdom | 63 | 61 | 124
  Czech Republic | 48 | 50 | 98
  Hungary | 17 | 19 | 36
  Mexico | 60 | 59 | 119
  Belgium | 27 | 25 | 52
  Brazil | 17 | 17 | 34
  Poland | 41 | 45 | 86
  Singapore | 8 | 9 | 17
  Norway | 35 | 36 | 71
  Germany | 122 | 122 | 244
  Sweden | 1 | 0 | 1
Type of Risk Factor [Number; unit: Participants]
  Knee replacement | 257 | 286 | 543
  Hip replacement | 90 | 80 | 170
  Hip or knee fracture surgery | 55 | 49 | 104
  Deep vein thrombosis | 36 | 32 | 68
  Pulmonary embolism | 10 | 10 | 20

OUTCOME MEASURES:

1. Secondary Outcome: Rate of Adjudicated Proximal Deep Vein Thrombosis (DVT), Nonfatal Pulmonary Embolism, and Venous Thromboembolic Event-related Death With Onset During the Intended Treatment Period
Description: Event rate=Number of events divided by the number of patients evaluated. Intended treatment period starts on the day of randomization, and for those who received study drug, ends at the later of 2 days after last dose or 14 days after the first dose of study drug; for randomized patients who did not receive study drug, the period ends 14 days after randomization; for randomized patients who did not receive study drug, the period ends 14 days after randomization. Venous thromboembolic event (VTE)=nonfatal pulmonary embolism (PE), symptomatic DVT, or asymptomatic proximal DVT detected by ultrasound. VTE-related death=fatal PE or sudden death for which VTE could not be excluded as a cause.
Time Frame: Day of randomization to later of 2 days after last dose or 14 days after first dose; 14 days after randomization for those who did not receive study
Population: Randomized participants with either an adjudicated and evaluable bilateral proximal venogram or an adjudicated event associated with the endpoint, during the Intended Treatment Period
Measure: Number (95% Confidence Interval); unit: Percentage of events/patients evaluated
Arm/Group | Apixaban, 2.5 mg BID + Placebo | Enoxaparin, 40 mg QD + Placebo
Number analyzed (Participants) | 1195 | 1199
Percentage of events/patients evaluated | 1.09 [0.62 to 1.88] | 2.17 [1.47 to 3.18]
Statistical Analysis 1: Comparison: Apixaban, 2.5 mg BID + Placebo vs Enoxaparin, 40 mg QD + Placebo; Sequential testing was used to control for overall type-I error and to compare the effect of apixaban with that of enoxaparin. Noninferiority (NI) of apixaban compared with enoxaparin for primary endpoint was tested first at 1-sided α=0.025 level. If superiority was demonstrated on the primary endpoint, NI was then tested on the secondary endpoint at a 1-sided α=0.025 level. If NI of the secondary endpoint was demonstrated, superiority was then tested at the 1-sided α=0.025 level; Test type: Superiority or Other; p = 0.0003, Yanagawa, Tango, and Hiejima test — 1-sided P-value; Risk Ratio (RR) = .50 — Apixaban-enoxaparin
Statistical Analysis 2: Comparison: Apixaban, 2.5 mg BID + Placebo vs Enoxaparin, 40 mg QD + Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Inverse variance method; Risk Difference (RD) = -1.04, 95% CI [-2.03 to -0.05]

2. Secondary Outcome: Rate of Major Bleeding, Clinically Relevant Nonmajor Bleeding (CRNM), and Major Bleeding or CRNM
Description: Event rate=Number of events divided by number of patients evaluated. Adjusted difference of event rates takes into consideration type of surgery as a stratification factor. Bleeding Criteria: Major bleeding=an event consisting of clinically overt bleeding accompanied by a decrease in hemoglobin of 2 g/dL or more and/or a transfusion of 2 or more units of packed red blood cells; bleeding that occurred in at least 1 of the following critical sites: intracranial, intraspinal, intraocular (within the corpus of the eye; a conjunctival bleed is not an intraocular bleed), pericardial, intra-articular, intramuscular with compartment syndrome, and retroperitoneal; bleeding that was fatal. CRNM bleeding= clinically overt bleeding; that satisfies none of the additional criteria required for the event to be adjudicated as a major bleeding event; that led to either hospital admission for bleeding, physician-guided medical or surgical treatment for bleeding; or a change in antithrombic treatment.
Time Frame: Days 1 to 12
Population: All participants who received at least 1 dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of events/patients evaluated
Arm/Group | Apixaban, 2.5 mg BID + Placebo | Enoxaparin, 40 mg QD + Placebo
Number analyzed (Participants) | 1501 | 1508
Percentage of events/patients evaluated
  Major bleeding (n=9, 14) | 0.60 [0.30 to 1.16] | 0.93 [0.54 to 1.57]
  CRNM (n=44, 58) | 2.93 [2.19 to 3.93] | 3.85 [2.98 to 4.95]
  Major bleeding or CRNM (n=53, 72) | 3.53 [2.71 to 4.60] | 4.77 [3.81 to 5.98]
  Any bleeding | 6.93 [5.75 to 8.34] | 8.36 [7.06 to 9.87]
Statistical Analysis 1: Comparison: Apixaban, 2.5 mg BID + Placebo vs Enoxaparin, 40 mg QD + Placebo; Major bleeding; Test type: Superiority or Other; p = 0.3014, Mantel Haenszel; Adjusted difference of event rates = -0.33, 95% CI 2-sided [-0.95 to 0.29] — Apixaban-enoxaparin
Statistical Analysis 2: Comparison: Apixaban, 2.5 mg BID + Placebo vs Enoxaparin, 40 mg QD + Placebo; CRNM; Test type: Superiority or Other; p = 0.1668, Mantel Haenszel; Adjusted difference of event rates = -0.91, 95% CI 2-sided [-2.20 to 0.38] — Apixaban-enoxaparin
Statistical Analysis 3: Comparison: Apixaban, 2.5 mg BID + Placebo vs Enoxaparin, 40 mg QD + Placebo; Major or CRNM; Test type: Superiority or Other; p = 0.0881, Mantel Haenszel; Adjusted difference of event rates = -1.24, 95% CI 2-sided [-2.66 to 0.18] — Apixaban-enoxaparin
Statistical Analysis 4: Comparison: Apixaban, 2.5 mg BID + Placebo vs Enoxaparin, 40 mg QD + Placebo; Any bleeding; Test type: Superiority or Other; p = 0.1412, Mantel Haenszel; Adjusted difference of event rates = -1.39, 95% CI 2-sided [-3.29 to 0.51] — Apixaban-enoxaparin

3. Primary Outcome: Rate of Adjudicated Venous Thromboembolic Event-related and All-cause Deaths With Onset During the Intended-treatment Period
Description: Event rate=Number of events divided by the number of patients evaluated. Intended treatment period starts on the day of randomization, and for those who received study drug, ends at the later of 2 days after last dose or 14 days after the first dose of study drug; for randomized patients who did not receive study drug, the period ends 14 days after randomization.Venous thromboembolic event (VTE)=nonfatal pulmonary embolism (PE), symptomatic deep vein thrombosis (DVT), or asymptomatic proximal DVT detected by ultrasound. VTE-related death=fatal PE or sudden death for which VTE could not be excluded as a cause.
Time Frame: Day of randomization to later of 2 days after last dose or 14 days after first dose; 14 days after randomization for those who did not receive study drug
Population: The primary efficacy data set (all randomized participants who, during the Intended Treatment Period, had an adjudicated and evaluable bilateral venogram, an adjudicated venous thrombolytic event; or died due to any cause.)
Measure: Number (95% Confidence Interval); unit: Percentage of events/patients evaluated
Groups:
- Apixaban, 2.5 mg BID: Participants received apixaban, 2.5 mg twice daily (BID), as oral tablets, and matching enoxaparin-placebo injection once daily (QD)
- Enoxaparin, 40 mg QD: Participants received enoxaparin, 40 mg QD subcutaneously, and matching apixaban-placebo tablets BID
Arm/Group | Apixaban, 2.5 mg BID | Enoxaparin, 40 mg QD
Number analyzed (Participants) | 976 | 997
Percentage of events/patients evaluated | 15.06 [12.95 to 17.46] | 24.37 [21.81 to 27.14]
Statistical Analysis 1: Comparison: Apixaban, 2.5 mg BID vs Enoxaparin, 40 mg QD; Sequential testing was used to control for overall type-I error and to compare the effect of apixaban with that of enoxaparin. Noninferiority (NI) of apixaban compared with enoxaparin for primary endpoint was tested first at 1-sided α=0.025 level. If NI on primary endpoint was demonstrated, superiority for the endpoint was then tested at 1-sided α=0.025 level. If superiority was demonstrated on the primary endpoint, NI was then tested on the key secondary endpoint at 1-sided α=0.025 level; Test type: Superiority or Other; p < 0.0001, Yanagawa, Tango, and Hiejima test — P-value was statistically significant at the 1-sided 0.025 level; Risk Ratio (RR) = 0.62, 95% CI 2-sided [0.51 to 0.74] — Apixaban-enoxaparin
Statistical Analysis 2: Comparison: Apixaban, 2.5 mg BID vs Enoxaparin, 40 mg QD; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.0001, Yanagawa, Tango, and Hiejima test — P-value is statistically significant at the 1-sided 0.025 level; Risk Difference (RD) = -9.27, 95% CI [-12.74 to -5.79] — Apixaban-enoxaparin

4. Secondary Outcome: Number of Participants With Serious Adverse Events (SAE), Bleeding Adverse Events (AEs), Discontinuations Due to AEs, and Death as Outcome
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Bleeding AEs=all serious or nonserious bleeding-related AEs.
Time Frame: Days 1 through 12 + 2 days (nonserious AEs, bleeding AES) or 30 days (SAES, deaths) after last dose of study drug
Population: All participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Apixaban, 2.5 mg BID + Placebo | Enoxaparin, 40 mg QD + Placebo
Number analyzed (Participants) | 1501 | 1508
Participants
  SAE | 72 | 88
  Bleeding AE | 90 | 112
  Discontinuations due to AEs | 40 | 44
  Deaths | 2 | 0

5. Other Pre Specified Outcome: Summary of Laboratory Marked Abnormalities on Hematology and Liver and Kidney Function Test Results During the Treatment Period (Patients With Available Measurements)
Description: preRX=pretreatment; LLN=lower limit of normal; ULN=upper limit of normal; abs=absolute. Hemoglobin (g/dL): >2 decrease from preRx value or value <=8; hematocrit (%): <0.75*preRx; platelets: <100*10^9 cells/L; erythrocytes (*10^6 cells/μL): <0.75*preRx; leukocytes: <0.75*LLN or >1.25*ULN, or if preRx <LLN, use <0.8*preRx or >ULN if preRx >ULN use >1.2*preRx or <LLN; abs basophils: >400/mm^3; abs eosinophils: > 0.750*10^3 cells/µL; abs lymphocytes: <0.750*10*3 cells/ µL or >7.50*10^3 c/ µL; abs monocytes > 2000/mm^3; abs neutrophils: <1.0*10^3 cells/μL; ALP (U/L): >2*ULN; ALT, AST (U/L): >3*ULN; U/L; bilirubin, direct (mg/dL): >1.5*ULN; bilirubin, total (mg/dL): >2*ULN; BUN (mg/dL): >2*ULN; creatinine (mg/dL): >1.5*ULN.
Time Frame: Randomization to Days 2, 3, 4, and 12 (±2 days) and at Days 42 and 72 (±5 days) of follow-up
Population: All participants who received at least 1 dose of study drug. n=number of participants with available measurements
Measure: Number; unit: Participants
Arm/Group | Apixaban, 2.5 mg BID + Placebo | Enoxaparin, 40 mg QD + Placebo
Number analyzed (Participants) | 1501 | 1508
Participants
  Hemoglobin, low (n=1424, 1442) | 1127 | 1178
  Hematocrit, low n=(1369, 1396) | 668 | 723
  Platelet count, low (n=1413, 1425) | 7 | 5
  Erythrocytes, low (n=1368, 1396) | 690 | 735
  Leukocytes, low (n=1457, 1471) | 27 | 26
  Leukocytes, high (n=1457, 1471) | 193 | 213
  Basophils (absolute), high (n=1448, 1465) | 2 | 4
  Eosinophils (absolute), high (n=1448, 1465) | 43 | 60
  Lymphocytes (absolute), low (n=1448, 1465) | 203 | 215
  Lymphocytes (absolute), high (n=1448, 1465) | 1 | 0
  Monocytes (absolute), high (n=1448, 1465) | 5 | 2
  Neutrophils (absolute), low (n=1448, 1465) | 5 | 2
  Alkaline phosphatase (ALP), high (n=1465, 1476) | 15 | 31
  Alanine aminotransferase (ALT), high (n=1459,1472) | 32 | 26
  Aspartate aminotransferase (AST) , high (n=1459,14 | 34 | 26
  Bilirubin, direct (high) (n=1447,1457) | 87 | 76
  Bilirubin, total (high) (n=1461,1476) | 15 | 9
  Blood urea nitrogen (BUN) (high)(n=1447,1458) | 15 | 17
  Creatinine (high) (n=1447,1458) | 17 | 23

6. Other Pre Specified Outcome: Summary of Laboratory Marked Abnormalities in Electrolyte and Other Clinical Test Results During the Treatment Period (Patients With Available Measurements)
Description: preRX=pretreatment; LLN=lower limit of normal; ULN=upper limit of normal. Calcium, total (mg/dL): <0.8*LLN or >1.2*ULN, or if preRx<LLN use <0.75*preRx or >ULN if preRx >ULN use >1.25*preRx or <LLN; chloride, serum (mEq/L): <0.9*LLN or >1.1*ULN, or if preRx<LLN use <0.9*preRx or >ULN if preRx>ULN use >1.1*preRx or <LLN; bicarbonate (mEq/L): <0.75*LLN or >1.25*ULN, or if preRx < LLN use <0.75*preRx or >ULN if preRx >ULN use >1.25*preRx or < LLN; potassium, serum (mEq/L): <0.9* LLN or >1.1*ULN, or if preRx<LLN use <0.9 *preRx or >ULN if preRx>ULN use >1.1*preRx or <LLN; sodium, serum (mEq/L): <0.95*LLN or >1.05*ULN, or if preRx <LLN use <0.95*preRx or >ULN if preRx>ULN use >1.05*preRx or <LLN; protein, total (g/dL): <0.9*LLN or >1.1*ULN, or if preRx <LLN use 0.9*preRx or >ULN if preRx >ULN use 1.1*preRx or <LLN; CK (U/L): >5*ULN; uric acid (mg/dL): >1.5*ULN, or if preRx >ULN use >2*preRx; glucose, fasting serum (mg/dL): <0.8*LLN or >1.5*ULN, or if preRx <LLN use <0.8*preRx or >ULN.
Time Frame: Randomization to Days 2, 3, 4, and 12 (±2 days) and at Days 42 and 72 (±5 days) of follow-up
Population: All participants who received at least 1 dose of study drug. n=number of participants with available measurements
Measure: Number; unit: Participants
Arm/Group | Apixaban, 2.5 mg BID + Placebo | Enoxaparin, 40 mg QD + Placebo
Number analyzed (Participants) | 1501 | 1508
Participants
  Calcium, total (low) (n=1447, 1457) | 5 | 9
  Chloride, serum (low)(n=1442, 1454) | 1 | 0
  Bicarbonate (low) (n=1435, 1447) | 0 | 3
  Potassium, serum (low) (n=1438, 1453) | 38 | 41
  Potassium, serum (high)(n=1438, 1453) | 34 | 40
  Sodium, serum (low) (n=1442, 1454) | 5 | 10
  Sodium, serum (high) (n=1442, 1454) | 1 | 0
  Glucose, fasting serum (low) (n=715, 713) | 8 | 1
  Glucose, fasting serum (high) (n=715, 713) | 46 | 25
  Protein, total (low) (n=1447, 1457 | 223 | 243
  Creatine kinase (CK) (high) (n=1463, 1476) | 66 | 65
  Uric acid (high) (n=1446, 1458) | 1 | 2

7. Other Pre Specified Outcome: Summary of Laboratory Marked Abnormalities in Urinalysis Results During the Treatment Period-Treated Subjects With Available Measurements (Urinalysis)
Description: preRX=pretreatment. Blood, urine: If missing preRx use ≥2, or if value ≥4, or if preRx=0 or 0.5 use ≥2, or if preRx=1 use ≥3, or if preRx=2 or 3 use ≥4; glucose, urine: If missing preRx use ≥2, or if value ≥4, or if preRx=0 or 0.5 use ≥2, or if preRx=1 use ≥3, or if preRx=2 or 3 use ≥4; protein, urine: If missing preRx use ≥ 2, or if value ≥4, or if preRx=0 or 0.5 use ≥2, or if preRx=1 use ≥3, or if preRx=2 or 3 use ≥4; Red blood cells , urine: If missing preRx use ≥2, or if value ≥4, or if preRx=0 or 0.5 use ≥2, or if preRx=1 use ≥3, or if preRx=2 or 3 use ≥4; white blood cells, urine: If missing preRx use ≥2, or if value ≥4, or if preRx=0 or 0.5 use ≥2, or if preRx=1 use ≥3, or if preRx=2 or 3 use ≥4.
Time Frame: Randomization to Days 2, 3, 4, and 12 (±2 days) and at Days 42 and 72 (± 5 days) of follow-up
Population: All participants who received at least 1 dose of study drug. n=number of participants with available measurements
Measure: Number; unit: Participants
Arm/Group | Apixaban, 2.5 mg BID + Placebo | Enoxaparin, 40 mg QD + Placebo
Number analyzed (Participants) | 1501 | 1508
Participants
  Blood, urine (high) (n=1421, 1430) | 169 | 113
  Glucose, urine (high) (n=1421, 1429) | 160 | 154
  Protein, urine (high) (n=1421, 1430) | 60 | 89
  Red blood cells, urine (high) (n=441, 385) | 133 | 116
  White blood cells, urine (high)(n=441, 386) | 101 | 102

ADVERSE EVENTS:
Groups:
- Apixiban, 2.5 mg BID Plus Placebo: Participants received apixaban, 2.5 mg twice daily (BID), as oral tablets, and matching enoxaparin-placebo injection once daily (QD)
- Enoxaparin, 40 mg QD Plus Placebo: Participants received enoxaparin, 40 mg QD subcutaneously, and matching apixaban-placebo tablets BID
Arm/Group | Apixiban, 2.5 mg BID Plus Placebo | Enoxaparin, 40 mg QD Plus Placebo
Serious Adverse Events (participants affected / at risk) | 72/1501 | 88/1508
Other Adverse Events (participants affected / at risk) | 295/1501 | 342/1508
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apixiban, 2.5 mg BID Plus Placebo (N=1501) | Enoxaparin, 40 mg QD Plus Placebo (N=1508)
Creatinine renal clearance decreased (Investigations) | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Hypokinesia (Nervous system disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Suture related complication (Injury, poisoning and procedural complications) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 2
Hypertensive crisis (Vascular disorders) | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Oedema peripheral (General disorders) | 2 | 2
Subcutaneous abscess (Infections and infestations) | 1 | 0
Wound haemorrhage (Vascular disorders) | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0
Device dislocation (Injury, poisoning and procedural complications) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erysipelas (Infections and infestations) | 2 | 1
Foreign body trauma (Injury, poisoning and procedural complications) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Injection site extravasation (General disorders) | 1 | 0
Platelet count increased (Investigations) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Senile dementia (Nervous system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Varicose vein (Vascular disorders) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Body temperature increased (Investigations) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 2
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Respiratory tract infection viral (Infections and infestations) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 1
Arthritis bacterial (Infections and infestations) | 1 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1
Death (General disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Oxygen saturation decreased (Investigations) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural infection (Infections and infestations) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Wound sepsis (Infections and infestations) | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1
Catheter related complication (General disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 1
Haemorrhage (Vascular disorders) | 4 | 3
Hypotension (Vascular disorders) | 0 | 1
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Postoperative wound infection (Infections and infestations) | 3 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Tuberculosis (Infections and infestations) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 5
Faecaloma (Gastrointestinal disorders) | 0 | 1
Haematoma (Vascular disorders) | 0 | 2
Hepatic enzyme increased (Investigations) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Localised infection (Infections and infestations) | 0 | 2
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 11 | 22
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Hepatic ischaemia (Hepatobiliary disorders) | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 1
Multi-organ failure (General disorders) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound infection (Infections and infestations) | 2 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Apixiban, 2.5 mg BID Plus Placebo (N=1501) | Enoxaparin, 40 mg QD Plus Placebo (N=1508)
Constipation (Gastrointestinal disorders) | 73 | 77
Vomiting (Gastrointestinal disorders) | 77 | 88
Nausea (Gastrointestinal disorders) | 102 | 120
Deep vein thrombosis (Vascular disorders) | 92 | 130

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication